CLINICAL TRIAL: NCT06460337
Title: Comparative Effects of Modified Otago and Frenkel's Exercises on Balance, Motor Function, Fear of Fall, and Quality of Life in Geriatric Population
Brief Title: Comparative Effects of Modified Otago and Frenkel's Exercises in Geriatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/23/0277
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Geriatrics
Keywords: Balance; Elderly; Frail older adults; Health-related quality of life; Exercise; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: It will be a randomized clinical trial. Through the computerized table generator method of randomization, the selected individuals will be evenly divided into two groups, one undergoing Frenkel's exercises and the other modified Otago exercises.
Who Masked: Outcomes Assessor
Masking Description: It is a single-blinded study, where the researcher who will assess outcomes, will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Otago Exercises (Experimental): It is a series of 17 strength and balance exercises in addition to 30 minutes walk outside the home at the usual pace three times a week.
  Interventions: Other: Modified Otago exercises
- Frenkel's Exercises (Active Comparator): It consists of simple range of motion exercises performed in different positions, i.e., lying, sitting, stride-standing and standing. Exercises are performed slowly emphasizing coordination and precision.
  Interventions: Other: Frenkel's exercises

INTERVENTIONS:
Other: Modified Otago exercises — Participants will engage in modified Otago exercise sessions, either individually or in groups, for 45 minutes, thrice weekly over an 8-week period. The program entails moderate-intensity strengthening exercises targeting various muscle groups such as hip extensors, abductors, knee flexors and extensors, inner range quadriceps, ankle plantar flexors, and dorsiflexors, performed at 10 repetitions maximum (RM) with ankle cuff weights ranging from 0.5 to 1 kg. Additionally, balance exercises will be conducted, initially with support and gradually progressing to without support, including knee bends, backwards walking, sideways walking, tandem stance and walk, one leg stance, heel and toe walking, sit-to-stand, stair climbing, stepping over objects, and bending to pick up objects from the floor. Participants are also encouraged to walk outdoors at their usual pace for 30 minutes at least three times weekly.
  Arms: Modified Otago Exercises
Other: Frenkel's exercises — Frenkel's exercise regimen comprises a series of movements performed in lying, sitting, stride standing, and standing positions aimed at improving coordination and motor control. In the lying position, exercises include alternating hip and knee flexion/extensions, hip abduction/adduction, pedaling the lower limbs, and simultaneous movements of hips and knees. These are executed slowly to enhance coordination. In sitting, exercises involve leg stretching, hip flexion with knees flexed or straightened, and transitions from sitting to standing and back. Stride standing exercises focus on weight transfer and sideways walking, while standing exercises encompass walking on marked paths, trunk rotations, 360-degree turns, smaller arcs of hip abduction/adduction and flexion/extension, straight-line walking, and directional changes to simulate real-life obstacles. 3 sets comprising 10 repetitions are performed for each exercise, aiming for motor skill improvement and balance enhancement
  Arms: Frenkel's Exercises

SUMMARY:
The goal of this randomized clinical trial is to compare the effects of modified Otago and Frenkel's exercises on balance, motor function, fear of fall and quality of life in the geriatric population. The main questions it aims to answer are:

* How modified Otago and Frenkel's exercises affect balance, motor function, fear of fall and quality of life in the geriatric population?
* Is there any difference between the effects of these two exercises? Researchers will compare the effects of modified Otago and Frenkel's exercises to see which kind of exercise has superior effects on the mentioned outcomes.

Participants will be randomly divided into two groups who will perform their respective exercises for 45 minutes 3 days a week for 8 weeks. Outcomes will be evaluated at the baseline, 4th week and 8th week.

DETAILED DESCRIPTION:
Several recent studies highlight the efficacy of various exercise interventions, including modified Otago and Frenkel's exercises, in improving balance, quality of life, and fear of falling among the elderly population. Many studies have demonstrated that Otago exercises show significant improvements in balance, fear of falling, and quality of life. In 2022, a study determined the impact of home-based Otago exercises on balance, quality of life, and fear of falling in the elderly. A meta-analysis conducted in 2021 evaluated the impact of the Otago Exercise Program. on both actual and perceived balance in older adults. In 2018, effects of Otago exercises were studies in comparison to Tai Chi. Similarly, in 2022, a study investigated the impact of Frenkel exercises combined with Cawthorne-Cooksey on functional balance and the risk of falling in the elderly. Moreover, in a study conducted in 2018, researchers evaluated the effects of Frenkel's exercise on improving balance in elderly patients, comparing it with aerobic exercise (walking). , in 2017, a study was carried out to analyze the effect of Frenkel's Exercises Vs. Swiss ball exercises on balance in patients with type II diabetic neuropathy. However, comparative research directly contrasting the effects of Otago and Frenkel's exercises on balance, motor function, and quality of life remains limited. Moreover, limited studies have explored the effects of Frenkel's exercises specifically on balance enhancement, emphasizing the need for further research in this area. Additionally, recent literature lacks detailed protocols for Otago exercises or modified Otago exercises, hindering the development of evidence-based recommendations tailored to the unique needs of older adults. This research underscores the importance of addressing this gap to optimize exercise strategies for promoting health and well-being in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults of both genders who have experienced a fall at least once in the previous year
* Minimum Berg Balance score of >40
* Able to independently walk and perform everyday activities without any walking aid

Exclusion Criteria:

* Unable to walk independently.
* Previous surgeries related to knee or hip joint replacement.
* Severe comorbidities such as stroke, unstable coronary artery disease, Parkinson's disease, and epilepsy.
* Patients with mental illness such as schizophrenia, dementia, and Alzheimer's disease
* Uncorrected visual, auditory, or vestibular impairments
* Having limb defects or any physical disability that prevents performing the exercises

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Mini-Best Test | 8th week
  Mini-BESTest (Balance Evaluation Systems Test) is a brief yet comprehensive clinical assessment designed to evaluate balance, mobility, and fall risk in older adults. Consisting of 14 items, it covers a range of balance-related functions such as anticipatory and reactive postural adjustments, sensory orientation, and dynamic gait movements. Each item is scored from 0 to 2, with higher scores indicating better performance, and the maximum achievable score is 28 points
Falls Efficacy Scale- International | 8th week
  The Falls Efficacy Scale-International (FES-I) is a 16-item self-report questionnaire designed to assess an individual's fear of falling during daily activities. Scores range from 16 to 64, with higher scores indicating greater fear of falling. Healthcare professionals commonly use the FES-I to identify individuals at risk of falling and to tailor interventions that improve confidence and reduce the fear of falling.
Older People's Quality of Life Questionnaire (OPQOL) | 8th week
  The Older People's Quality of Life Questionnaire (OPQOL) is a self-report tool designed to assess the multidimensional aspects of well-being in older adults. Covering domains such as physical health, psychological well-being, social relationships, and overall life satisfaction, the OPQOL provides a comprehensive understanding of the quality of life for older individuals. It consists of 35 questions with answers on 5-point Likert scale. The total score can range from 35 to 175, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (1):
- Wahla Family Hospital, Pindi Bhattian, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jahanpeyma P, Kayhan Kocak FO, Yildirim Y, Sahin S, Senuzun Aykar F. Effects of the Otago exercise program on falls, balance, and physical performance in older nursing home residents with high fall risk: a randomized controlled trial. Eur Geriatr Med. 2021 Feb;12(1):107-115. doi: 10.1007/s41999-020-00403-1. Epub 2020 Nov 25. PMID 33237565
- [Background] Manko G, Pieniazek M, Tim S, Jekielek M. The Effect of Frankel's Stabilization Exercises and Stabilometric Platform in the Balance in Elderly Patients: A Randomized Clinical Trial. Medicina (Kaunas). 2019 Sep 11;55(9):583. doi: 10.3390/medicina55090583. PMID 31514453